CLINICAL TRIAL: NCT06536543
Title: Pulmonary Overdistension Assessment With Electrical Impedance Tomography in Patients With Acute Respiratory Distress Syndrom in Prone Position
Brief Title: EIT Assessment of Overdistension in ARDS Patients in Prone Position
Acronym: DISTIE-DV
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2022/13
Record Dates: First submitted 2024-07-26; First posted 2024-08-05 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: Ventilation Induced Lung Injury; lung overdistension; lung collapse; Electrical Impedance Tomography; Pressure Volume curve; Prone Position
MeSH Terms: conditions — Respiratory Distress Syndrome; Pulmonary Atelectasis | interventions — Therapeutics; Prone Position

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Patients with moderate or severe ARDS treated with PP equipped with EIT will be included.
  Measurement of EIT data and ventilator spirometry in supine position and just after turning the patient in PP during a decremental PEEP-EIT titration, will be done, and blood gases and finally haemodynamic data
  Interventions: Other: Acute Respiratory Distress Syndrom (ARDS) treated with Prone Position (PP) equipped with Electrical Impedance Tomography (EIT)

INTERVENTIONS:
Other: Acute Respiratory Distress Syndrom (ARDS) treated with Prone Position (PP) equipped with Electrical Impedance Tomography (EIT) — Positive End-Expiratory Pressure (PEEP) will be titrated with PEEP-EIT method as it is already done in usual care. A classical low flow Pression Volume (PV) curve will be done in order to detect airway closure and measure compliance, the acquisition of EIT data during PV curve will be analysed secondary with a dedicated software. Reconstruction of EIT derived PV curve will determine the regional airway opening pressures and compliances of the 2 lungs. Two decremental PEEP-EIT titrations will be compared, one in supine and the other just after turning in prone.

SUMMARY:
Mechanical ventilation in ARDS requires protective ventilation with low VT and PEEP. PEEP titration can improve lung recruitment in the dependent lung but with a risk of overdistension in the non-dependant lung. EIT can measure the distribution of tidal ventilation and assess overdistension and collapse during a PEEP titration in any position (prone or not).

This study aims to measure the best PEEP as a compromise between recruitment and overdistension during a PEEP trial with EIT before and just after PP.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized in the ICU and who suffered moderate or severe ARDS (Berlin criteria, PaO2/FiO2<150), intubated sedated, under myorelaxant and equipped with EIT
* Over the age of 18.

Exclusion Criteria:

* Broncho-pleural leaks
* Pregnant or breastfeeding woman.
* Guardianship or curatorship
* Deprived of liberty
* No health insurance
* Impossibility to correctly position the EIT belt (e.g., dressings, chest drainage, etc.)
* Contra indications to EIT (e.g., implantable cardiac defibrillator, pacemaker, instable spinal lesions)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalised in the thoracic intensive care unit, with moderate or severe ARDS according to the Berlin criteria, requiring a prone position, treated with PP equipped with EIT, will be included.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Level of distension | 48 hours after inclusion day
  Assessing the level of distension when titrating the optimal PEEP in the supine position (SP) and in the PP position the first and second day of ARDS in PP. The measure will be obtained thanks to the crossing in EIT of the overdistension curve and the collapse curve when the PEEP is reduced from 20 to 5 cmH2O.

SECONDARY OUTCOMES:
Comparison of the percent of overdistension and collapse during the EIT-PEEP titration | 48 hours after inclusion day
  Thanks to PEEP-EIT titration in PP and SP the percent of collapse and global over-distension in EIT will be evaluate.
Repartition of regional ventilation in each part of the lungs. | 48 hours after inclusion day
  Thanks to PV-EIT curve, the measurement of regional Airway Opening Pressure (anterior vs posterior) will be evaluate (lower inflection point of the PV-EIT curve).

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CH Cote Basque, Bayonne
  - Hopital Haut-Lévêque, Pessac